CLINICAL TRIAL: NCT00488449
Title: A Two-Part Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Oral Doses of GSK256073A, in a Randomized, Single-Blind, Dose Escalation Study in Healthy Adult Subjects
Brief Title: Study Of Pharmacokinetics and Pharmacodynamics Effects Of GSK256073A On Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HMA110015
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Dyslipidaemias
Keywords: Dose Escalation; GSK256073A,

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256073A tablets

SUMMARY:
The purpose of this study is to compare the effects of single and repeat doses of GSK256073 with placebo in HVT subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy Adult males or females between 18 and 55 years of age, inclusive.
* Female subjects must be of non-childbearing potential
* Body weight > 50 kg (110 pounds) and body mass index (BMI) 19 and 31 where:
* Subjects with QTc < 450 msec at screening (or QTc < 480 msec for subjects with Bundle Branch Block).
* A signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restriction

Exclusion criteria:

* Systolic blood pressure < 100 mmHg or 150 mmHg and/or diastolic blood pressure = 100 mmHg at screening.
* History of significant cardiac arrhythmias
* Active peptic ulcer disease (PUD) and/or history of PUD within 1 year.
* A serum uric acid concentration 8mg/dL
* Screening test positive for H. Pylori using the non-radioactive breath test
* History of gout and/or hyperuricemia
* History of Gilbert's syndrome
* A serum creatinine concentration above the normal reference range
* History of kidney stones
* PT and/or aPTT above the reference range
* History of recurrent indigestion, stomach upset or diarrhea
* Liver function tests (LFTs) or creatinine phosphokinase (CPK) 1.5X ULN
* Screening stool test positive for occult blood
* Screening peripheral blood smear with abnormal RBCs
* CBC, MCV, and/or reticulocyte count corrected for haemoglobin level above the reference range at screening
* Reduced G6PD activity
* Serum haptoglobin outside the reference range at screening
* Total serum LDH > 1.25% above the ULN at screening
* Positive HIV, Hepatitis B or Hepatitis C at screening
* The subject has a positive pre-study urine drug/ serum alcohol screen.
* History of alcohol consumption exceeding, on average, 7 drinks/week for women or 14 drinks/week for men within 6 months of the first dose of study medication or a positive alcohol test at screening
* History of use of tobacco or nicotine containing products within 6 months of screening or a positive urine cotinine screen
* Use of prescription (including hormone replacement therapy) or non-prescription drugs and vitamins within 7 days or 5 half-lives prior to administration of study medication. An exception is acetaminophen which is allowed at doses of 2g/day.
* Use of dietary/herbal supplements within 14 days prior to treatment with study medication
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.
* Unwillingness of male subjects to use a condom/spermicide
* Pregnant or nursing women.
* History of flushing (>1 episode annually).
* Fasting blood glucose 110 mg/dl and/or history of type I or type II DM
* History of intra-ocular pathology
* History of recurrent gum bleeding
* History of bleeding haemorrhoids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
AEs, 12-Lead ECG, vital signs, nursing/physician observation, safety lab tests, flushing | throughout the study (Parts A &B)
AUC and Cmax | throughout the study (Part A & B)
Measures of accumulation ratios | throughout the study (Ro, Rp, and Rs)[Part B]

SECONDARY OUTCOMES:
Tmax, t½, Ae, and CLr (Parts A & B) Cmax, ss, Ct, t½, Ae, CLr, and accumulation ratios (Part B) | throughout the study
PD response: NEFA and TG (6 and 24 hours post- dose) | (6 and 24 hours post- dose)
LDL, HDL, ApoA1, ApoA2, Apo B and Lp(a) | on Days 1, 14, and 15.
Levels of GSK256073 to derive pharmacokinetic parameters following repeat dose administration.
Lipid levels | on Days 1, 14, and 15

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States